CLINICAL TRIAL: NCT03180190
Title: Cytochrome P450 and ATP-Binding Cassette C C (ABCC) Variants in Egyptian Patients Receiving Hydroxychloroquine and Their Association With Efficacy and Toxicity
Brief Title: Genetic Variants in Egyptian Patients Receiving HCQ(Hydroxychloroquine)
Acronym: HCQ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, nesreen ismail ibrahim, principle investigator, Assiut University
Other Study IDs: Hydroxychloroquine
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — Hydroxychloroquine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — 5 ml of blood will be collected into tubes containing EDTA, and stored immediately at -80 for genomic DNA extraction and genotyping using real time PCR (Taqman discrimination assay) for study frequency of single nucleotide polymorphisms (SNPs)of CYP2C19, CYP1A2, and ABCG2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with ocular toxicity: Screening for ophthalmic exclusion criteria by slit lamp and fundus examination using both direct and indirect ophthalmoscope Screening for HCQ ocular toxicity by
  * Perimetry using Octopus perimeter and utilizing 24-2 test strategy,
  * Electroretinography (ERG) under scotopic and photopic conditions and Spectral domain optical coherence tomography (SD-OCT) genotyping using real time PCR (Taqman discrimination assay) for study frequency of single nucleotide polymorphisms (SNPs) of CYP2C19, CYP1A2, and ABCG2.
  Interventions: Drug: Hydroxychloroquine Oral Tablet
- patients without ocular toxicity: Screening for ophthalmic exclusion criteria by slit lamp and fundus examination using both direct and indirect ophthalmoscope Screening for HCQ ocular toxicity by
  * Perimetry using Octopus perimeter and utilizing 24-2 test strategy,
  * Electroretinography (ERG) under scotopic and photopic conditions and Spectral domain optical coherence tomography (SD-OCT) genotyping using real time PCR (Taqman discrimination assay) for study frequency of single nucleotide polymorphisms (SNPs) of CYP2C19, CYP1A2, and ABCG2.
  Interventions: Drug: Hydroxychloroquine Oral Tablet

INTERVENTIONS:
Drug: Hydroxychloroquine Oral Tablet — slit lamp and fundus examination using both direct and indirect ophthalmoscope Screening for HCQ ocular toxicity by
  * Perimetry using Octopus perimeter and utilizing 24-2 test strategy,
  * Electroretinography (ERG) under scotopic and photopic conditions and Spectral domain optical coherence tomography (SD-OCT)
  Other Names: diagnostic test

SUMMARY:
Hydroxychloroquine(HCQ)play major role in management of many rheumatic diseases.

Retinal toxicity from HCQ is serious side effect because even after the drug drug is discontinued, there is little if any visual recovery. For this reason, regular screening for retinal toxicity is recommended to detect early retinopathy and discontinue the therapy.

Cytochrome P450 (CYP) enzymes play major roles in drug metabolism. Certain single-nucleotide polymorphisms(SNPs) in CYP genes may have a large impact on CYP enzyme activity.Polymorphisms in the cytochrome P450 gene might influence blood concentration some patients have a genetic predisposition to HCQ toxicity (e.g.,from abnormalities in the ABCA4 gene)Which is not studied previously among Egyptian population

DETAILED DESCRIPTION:
The antimalarial agent hydroxychloroquine have been used widely for the treatment of rheumatoid arthritis and systemic lupus erythematosus.

Among rheumatic diseases, the primary role of HCQ is in the management of articular and skin manifestations of systemic lupus erythematosus (SLE) and the treatment of mild to moderately active rheumatoid arthritis (RA). As a cornerstone of SLE management, HCQ leads to reduction in the risk of disease flare as well as providing a valuable adjunct in the therapy of lupus nephritis, and is a relatively safe option for t0reatment of SLE during pregnancy,It also has been linked to the prevention thrombosis as well as a reduced risk of permanent organ damage. HCQ's beneficial effects on lipid levels and reduction in the risk of diabetes .It is a member of the "triple therapy" triad for the treatment of RA , serving as an important component of the therapeutic approach in active disease. Other less common uses for HCQ include the treatment of palindromic rheumatism, Inflammatory cutaneous disorders, and the antiphospholipid antibody syndrome because of its antithrombotic effect .

Retinal toxicity from HCQ is of serious ophthalmologic concern. Because even after the drug is discontinued, there is little if any visual recovery. Additionally, it has been shown that the retinal degeneration caused by HCQ can continue to progress. For this reason, regular screening for retinal toxicity is recommended to detect early retinopathy and discontinue the therapy.

The exact mechanism of HCQ and CQ toxicity remains unclear. Previously, it was hypothesized that retinal toxicity results from binding of HCQ and CQ to melanin in the retinal pigment epithelium (RPE), thus damaging the overlying photoreceptors and ultimately causing vision loss .Whether the primary effect of antimalarials occurs at the level of the RPE versus the retinal photoreceptors has been debated, however, as newer imaging technology has become available ,Early retinal toxicity is generally asymptomatic, with subtle alterations in foveal pigmentation that are often not evident on routine ophthalmologic examination. As toxicity progresses, classic "bull's eye" maculopathy, representing a ring of parafoveal RPE depigmentation sparing the central fovea, may be noted. Progression leads to increasing visual impairment, symptomatically manifesting as decreased central vision, reduced color vision, reduced night vision, reading difficulties, central scotomata, flashing lights, and increasing visual field defects.

Cytochrome P450 (CYP) enzymes play major roles in drug metabolism. Certain single-nucleotide polymorphisms(SNPs) in CYP genes may have a large impact on CYP enzyme activity.Polymorphisms in the cytochrome P450 gene might influence blood concentration.

HCQ is metabolized to N-desethyl HCQ (DHCQ) in the liver through the N-desethylation pathway,This reaction is mediated by CYP 2D6, 3A4, 3A5, and 2C8 isoforms.

some patients have a genetic predisposition to HCQ toxicity (e.g.,from abnormalities in the ABCA4 gene) However, in 2015 ABCA4 polymorphisms proposed that could be protective agent. Which is not studied previously among Egyptian population

ELIGIBILITY:
Inclusion Criteria:

* All patients received HCQ treatment and attending the Rheumatology and Rehabilitation outpatient clinic and in-patient department, Faculty of Medicine, Assiut University Hospitals.

Exclusion Criteria:

* • Patients less than 18 years old.

  * Patients with co-morbidities (e.g., liver disease, serious infections, or cardiac, respiratory, gastrointestinal, endocrine disease) that could influence the disease activity and the liver condition.
  * Patients with Renal failure (creatinine clearance < 30 ml/ min).
  * Patients with ophthalmic conditions that may give rise to abnormalities in the screening tests used to detect HCQ toxicity e.g. glaucoma, hereditary fundus dystrophies, dense media opacity precluding fundus visibility, optic neuritis and uveitis.
  * Patients receiving tamoxifen or other retinal toxin drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients receiving HCQ treatment
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-28 (Estimated); Primary Completion 2018-06-28 (Estimated); Study Completion 2018-07-28 (Estimated)

PRIMARY OUTCOMES:
HCQ toxicity in Egyptian patients | 1 year
  Recognizing clinical and genetic factor(s) affecting the outcome of HCQ therapy in Egyptian patients population and /or predisposing to its toxicity.

SECONDARY OUTCOMES:
genetic variant | 1 year
  Detecting the frequency (distribution) of single nucleotide polymorphisms (SNPs) of CYP and ABCC in Egyptian patients

IPD SHARING:
Plan to Share IPD: No